CLINICAL TRIAL: NCT01947257
Title: Is There a Correlation Between the Pulmonary Artery Pressure and the Acceleration of the Flow in the Pulmonary Artery Evaluated by Transesophageal Echocardiography (TOE) ?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-A00730-45; 2013-19 (Other: AP HM)
Record Dates: First submitted 2013-07-31; First posted 2013-09-20 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Ventilated Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ventilated patients (Other)
  Interventions: Other: the measure TRVMAX; Other: the measure of the pulmonary artery; Other: the direct measure of the pulmonary pressures

INTERVENTIONS:
Other: the measure TRVMAX — by transthoracic echocardiography
Other: the measure of the pulmonary artery — by transesophageal ultrasound
Other: the direct measure of the pulmonary pressures — by right catheterization

SUMMARY:
The measure of the pulmonary artery pressure (PAP) is a very useful index in intensive care to estimate right ventricular after load. The reference technique for this measure is the right catheterism which is an invasive technique. It is possible to estimate the pulmonary artery pressure by using transthoracic echocardiography (TTE) which allows, using the continuous Doppler, the measure of maximum speed of tricuspid regurgitation (TRvmax). The measure of the TRvmax can however be difficult for intensive care patients with little echogenicity or impossible for those having no tricuspid leak. The evaluation of the tricuspid regurgitation is also particularly difficult using TOE. To avoid these drawbacks, one can use the analysis of the pulmonary ejection in the pulmonary artery (PAAT) with TOE. However, the data of the literature are controversial on this method and it was not validated in mechanically ventilated intensive care patients.

The aim of this work is to compare three methods of measure of the PAP: the measure TRVMAX (by means of the tricuspid leak) by transthoracic echocardiography, the measure of the TAAP by transesophageal ultrasound and the direct measure of the pulmonary pressures by right catheterization, in ventilated patients already monitored with a catheter in the right cavities for usual indications in intensive care (ARDS, shock). We shall analyze then the correlation between the TRVmax, the TAAP and the pressures measured by the right catheterism which serves as reference technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Admitted to intensive care
* Mechanically ventilated and sedated
* Carrying a right catheterization
* Making a ETO indicated by the medical team or doctor in charge of the patient

Exclusion Criteria:

* Patients under 18 years
* expectant mother
* Patients without health insurance
* Refusal to close

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
measure of the pulmonary artery pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France